CLINICAL TRIAL: NCT00903929
Title: Phase I Study of Eltrombopag for Promoting Thrombopoiesis in Patients Undergoing Stem Cell Transplantation After Total Body Irradiation
Brief Title: Phase I Study of Eltrombopag for Promoting Thrombopoiesis After Total Body Irradiation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jane Liesveld (Other)
Responsible Party: Sponsor-Investigator, Jane Liesveld, Professor M&D-Hematology/Oncology, University of Rochester
Organization: University of Rochester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSRB00028043
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Results first posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-04

CONDITIONS: Thrombocytopenia; Acute Radiation Syndrome
MeSH Terms: conditions — Thrombocytopenia; Acute Radiation Syndrome | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eltrombopag (Experimental)
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — dose escalation

SUMMARY:
Patients who undergo total body irradiation (TBI) for stem cell transplantation have prolonged periods of low counts of specific blood cells called platelets. These low platelets counts can cause bleeding and infection. Thus far, no drug is available for use to speed the recovery of platelets, and therefore transfusions are often necessary.

The purpose of this study is to test the safety of a drug called eltrombopag in patients who have received TBI. The investigators want to find out what effects, good or bad, it has on people with low platelet counts due to treatment with TBI. The investigators will also be testing how well eltrombopag may work at different doses and determine if this drug speeds up the recovery of the platelets.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. Able to give written informed consent for a clinical trial
3. Scheduled to undergo an autologous or an allogeneic stem cell transplantation from a sibling, related donor, or unrelated donor using a conditioning regimen containing at least 400 cGy TBI
4. Transplantation is being performed for one of the following medical conditions:

   * Acute myelogenous leukemia
   * Acute lymphoblastic leukemia
   * Chronic myelogenous leukemia in chronic, accelerated, or blastic phase
   * Myelodysplastic syndrome
   * Myeloproliferative diseases such as chronic myelomonocytic leukemia, agnogeneic myeloid metaplasia with myelofibrosis, polycythemia vera, or essential thrombocythemia
   * Hodgkin's lymphoma
   * Non-Hodgkin's lymphoma
   * Multiple myeloma
   * Chronic lymphocytic leukemia
   * Other malignancies or marrow disease such as aplastic anemia where transplant would be appropriate with approval of principal investigator
5. Patients with therapy-related AML or MDS may be included if their prior malignancy has been in remission for at least 12 months. If the remission is less than 12 months, approval of the principal investigator is required. Entry could be allowed if the malignancy is controlled and not expected to relapse e.g. localized prostate cancer treated with XRT.
6. Patients must meet all other pre-transplantation criteria of the transplant center including acceptable tests of heart, liver, kidney, and lung function (Standard screening for HSCT per PI, and co-investigators).
7. Karnofsky performance status must be ≥70%.

Exclusion Criteria:

1. TBI dose less than 400 cGY
2. Cord blood transplantation
3. HIV infection
4. Pregnancy or breastfeeding
5. Creatinine or bilirubin or ALT or AST greater than two times the upper limit of normal, unless the abnormal bilirubin is due to Gilbert's syndrome
6. Active infection requiring systemic antibiotic therapy with antibacterial, antifungal, or antiviral agents
7. Concomitant enrollment in another therapeutic clinical study except with PI approval
8. Must not have previously received eltrombopag
9. Patients with moderate or severe liver disease (ALT, AST, or bilirubin ≥ 2X the upper limit of normal, unless the abnormal bilirubin is due to Gilbert's syndrome) will be excluded
10. Patients with high risk of thromboembolism based on genetic syndromes , or past thromboembolic disease in the past 6 months will be excluded from the study, with the exception of those with catheter related clots

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuhchyau Chen, MD,PhD, Study Director — University of Rochester; Jane Liesveld, MD, Principal Investigator — University of Rochester

REFERENCES:
- [Derived] Liesveld JL, Phillips GL 2nd, Becker M, Constine LS, Friedberg J, Andolina JR, Milner LA, DeBolt J, Smudzin T, Hyrien O, Erickson-Miller CL, Johnson BM, Dawson KL, Chen Y. A phase 1 trial of eltrombopag in patients undergoing stem cell transplantation after total body irradiation. Biol Blood Marrow Transplant. 2013 Dec;19(12):1745-52. doi: 10.1016/j.bbmt.2013.10.002. Epub 2013 Oct 8. PMID 24120380

RESULTS

PARTICIPANT FLOW:
Groups:
- Eltrombopag 75 mg; Eltrombopag 150 mg; Eltrombopag 225 mg; Eltrombopag 300 mg: Dose escalation was based on a standard 3+3 design. A group of 3 patients were enrolled at a given dose level; if none of these patients experienced dose-limiting toxicity (DLT), then the dose could be escalated. If 1 of the 3 patients experienced DLT, then 3 more patients would be enrolled at the same dose level. If no additional patients experienced a DLT, then dose escalation could occur, but if 2 or more of the 6 patients experienced a DLT, then that dose would be the MTD.
Period: Overall Study
Arm/Group | Eltrombopag 75 mg | Eltrombopag 150 mg | Eltrombopag 225 mg | Eltrombopag 300 mg
Started | 3 | 3 | 4 (Participants who did not complete the study were replaced with additional participants.) | 9 (Participants who did not complete the study were replaced with additional participants.)
Completed | 3 | 3 | 3 | 6
Not Completed | 0 | 0 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eltrombopag
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 52 [20 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Eltrombopag
Description: The MTD was defined as the highest dose if no dose limiting toxicity was observed, or the highest dose at which less than one-third of the patients experienced toxicities not expected in the standard stem cell transplantation setting.
Time Frame: 1.5 years
Measure: Number; unit: mg/day
Arm/Group | All Participants
Number analyzed (Participants) | 19
mg/day | 300

2. Secondary Outcome: Median Time to Platelet Engraftment
Description: Determined for all participants who completed at least 75% of the planned doses. Platelet engraftment was as defined by the Center for International Blood and Marrow Transplant Research as the first of 3 consecutive days of a platelet count 20,000/mL without platelet trans-fusions for 7 days and/or the first day of a platelet count 100,000/mL without platelet transfusions for 7 days.
Time Frame: 1.5 years
Measure: Median (Full Range); unit: days
Arm/Group | Eltrombopag
Number analyzed (Participants) | 19
days | 16 [0 to 86]

3. Secondary Outcome: Median Number of Platelet Transfusions up to the Day of Engraftment
Time Frame: baseline to day of engraftment
Measure: Median (Full Range); unit: units of platelets
Arm/Group | Eltrombopag
Number analyzed (Participants) | 19
units of platelets | 4 [0 to 68]

ADVERSE EVENTS:
Arm/Group | Eltrombopag
Serious Adverse Events (participants affected / at risk) | 8/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=19)
urosepsis (Infections and infestations) | 1
pumonary embolism (Vascular disorders) | 1
cytomegalovirus infection with fever (Infections and infestations) | 1
clostridium difficile infection (Infections and infestations) | 1
acute renal failure (Renal and urinary disorders) | 3
graft-versus-host disease of the gut (Gastrointestinal disorders) | 1
gastroparesis (Gastrointestinal disorders) | 1
acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
pericarditis (Cardiac disorders) | 1
graft-versus-host disease skin rash (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=19)
hypertension (Cardiac disorders) | 2
fatigue (General disorders) | 2
dehydration (Gastrointestinal disorders) | 2
diarrhea (Gastrointestinal disorders) | 3
dysphagia (Gastrointestinal disorders) | 3
mucositis (Gastrointestinal disorders) | 5
nausea (Gastrointestinal disorders) | 6
fever (Infections and infestations) | 6
infection with normal absolute neutrophil count (Infections and infestations) | 2
BK viruria (Infections and infestations) | 2
CMV reactivation (Infections and infestations) | 4
edema (Blood and lymphatic system disorders) | 3
hyperglycemia (Endocrine disorders) | 9
hypertriglyceridemia (Endocrine disorders) | 2
hypocalcemia (Endocrine disorders) | 2
hypomagnesemia (Endocrine disorders) | 2
hypokalemia (Endocrine disorders) | 5
hypophosphatemia (Endocrine disorders) | 3
syncope (Nervous system disorders) | 2
pain (Gastrointestinal disorders) | 3
headache (Nervous system disorders) | 4
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
hiccoughs (Respiratory, thoracic and mediastinal disorders) | 2
renal failure (Renal and urinary disorders) | 3
alanine aminotransferase elevation (Hepatobiliary disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes